CLINICAL TRIAL: NCT05668104
Title: Jing Si Herbal Tea Liquid Packet in the Treatment of Dyspeptic Symptoms and Psychophysical Burden in Patients With Disorders of Long-Coronavirus Disease(COVID) Gut-brain Interaction --a Double-blind, Randomized, Placebo Controlled Study
Brief Title: Jing Si Herbal Tea for Long-Coronavirus Disease(COVID) Gut-brain Interaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB111-232-A
Record Dates: First submitted 2022-12-26; First posted 2022-12-29 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2022-12

CONDITIONS: Healthy Subjects; COVID-19 Pneumonia; Irritable Bowel Syndrome; Functional Gastrointestinal Disorders
Keywords: functional dyspepsia; Jing Si Herbal Tea Liquid Packet; psychophysical burden; Gut-brain axis dysregulation
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jing Si Herbal Tea Liquid Packet (Experimental): Participants received Jing Si Herbal Tea Liquid Packet 15 mg tablet orally twice daily for 28 days.
  Interventions: Dietary Supplement: Jing Si Herbal Tea Liquid Packet
- Jing Si Herbal Tea Liquid Packet Placebo (Placebo Comparator): Participants received Jing Si Herbal Tea Liquid Packet Placebo 15 mg tablet orally twice daily for 28 days.
  Interventions: Dietary Supplement: Jing Si Herbal Tea Liquid Packet Placebo

INTERVENTIONS:
Dietary Supplement: Jing Si Herbal Tea Liquid Packet — The preliminary data demonstrated that the Jing Si Herbal Tea Liquid Packet may improve gastrointestinal symptoms and anxiety in patients with Coronavirus disease 2019(COVID-19). Therefore,this study aims to investigate the impact of the Jing Si Herbal Tea Liquid Packet on psychophysical burden and metabolites of microbiota in patients with FD through a double-blind randomized manner.
  Arms: Jing Si Herbal Tea Liquid Packet
Dietary Supplement: Jing Si Herbal Tea Liquid Packet Placebo — Compared with the improvement effect of Jing Si Herbal Tea Liquid Packet, to avoid participants thinking that the improvement is due to psychological effects.
  Other Names: Placebo
  Arms: Jing Si Herbal Tea Liquid Packet Placebo

SUMMARY:
Dyspepsia refers to chronic or recurrent upper gastrointestinal symptoms. According to the Rome IV criteria, functional dyspepsia (FD) symptoms included meal related fullness, early satiation, epigastric pain or burning which are unexpl ained after routine investigation. FD causes substantial psychophysical burden because of its unknown etiology and high prevalence. Although FD is currently associated with local inflammation of the gastrointestinal tract and microbiota alteration, current available treatments for FD are of limited effectiveness. In view of this, many studies have applied Chinese herbal medicine in FD and achieved some therapeutic benefit. The Jing Si Herbal Tea Liquid Packet composed of eight native Taiwanese herbs (wormwo od, hickory grass, Ophiopogon japonicus, houttuynia cordata, platycodon,licorice, perilla leaves, chrysanthemum) has obtained a special export license from the Ministry of Health and Welfare. The Jing Si Herbal Tea Liquid Packet also has been registered i n clinical trials as a complementary treatment for Coronavirus disease 2019(COVID-19). The preliminary data demonstrated that the Jing Si Herbal Tea Liquid Packet may improve gastrointestinal symptoms and anxiety in patients with COVID-19. Therefore,this study aims to investigate the impact of the Jing Si Herbal Tea Liquid Packet on psychophysical burden and metabolites of microbiota in patients with FD through a double blind randomized manner.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-70 years old.
2. Those who meet the definition of functional dyspepsia (FD). (Functional dyspepsia (FD) is chronic (once a week, lasting at least three months, at least six months before the first symptom) upper gastrointestinal symptoms (any of the following): postprandial abdominal distension, easy to feel full, Epigastric pain or burning sensation in the upper abdomen, and no symptoms of gastrointestinal bleeding or significant weight loss, no abnormality after upper gastrointestinal endoscopy).
3. Those who meet the definition of irritable bowel syndrome (IBS). (Irritable bowel syndrome (IBS) is chronic (once a week, lasting for at least three months) lower gastrointestinal symptoms: abdominal pain combined with diarrhea or constipation, and no symptoms of gastrointestinal bleeding or significant weight loss, no abnormalities after colonoscopy) .
4. Be conscious and willing to sign the subject's consent form.

Exclusion Criteria:

1. Abnormal liver and kidney function;
2. Abnormal blood tests and thyroid abnormalities;
3. Have received surgery on the digestive tract;
4. Abnormal upper gastrointestinal endoscopy;
5. Abnormal colonoscopy;
6. Antibiotics are being used for infectious diseases;
7. Pregnant or breastfeeding women;
8. Suffering from heart, liver, or kidney failure;
9. Physical weakness, allergies, asthenia and cold constitution and chronic diseases.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain on the Visual Analogue Scale (VAS) at day 28 | Baseline and day 28
  Possible scores range from 0 (No pain) to 10 (Worst possible pain) Change = (day 28 Score - Baseline Score).
Change from Baseline in Pain on the Gastrointestinal symptom rating scale (GSRS) at day 28 | Baseline and day 28
  Possible scores range from 1 (No pain) to 4 (Worst possible pain)
  1=No pain 2=Mild 3=Moderate 4=Worst possible pain Change = (day 28 Score - Baseline Score).
Change from Baseline on the Pittsburgh sleep quality index (PSQI) at day 28 | Baseline and day 28
  Possible scores range from 0 (Never) to 3 (Occurs three times a week times or more) 0=Never 1=Less than once a week 2=Occurs once or twice a week 3=Occurs three times a week times or more Change = (day 28 Score - Baseline Score).
Change from Baseline on the Taiwanese Depression Scale (TDQ) at day 28 | Baseline and day 28
  Possible scores range from 0 (Never) to 3 (Always) 0=Never 1=Sometimes 2=Often 3=Always Change = (day 28 Score - Baseline Score).
Change from Baseline on the State-Trait Anxiety Inventory (STAI) at day 28 | Baseline and day 28
  Possible scores range from 1 (Never) to 4 (Always)
  1=Never 2=Sometimes 3=Often 4=Always Change = (day 28 Score - Baseline Score).
Change from Baseline on the Perceived Stress Scale(PSS-10) at day 28 | Baseline and day 28
  Possible scores range from 0 (Never) to 4 (Always) 0=Never 1=Rarely 2=Sometimes 3=Often 4=Always Change = (day 28 Score - Baseline Score).
Change from Baseline on the Functional Dyspepsia Scale(FD) at day 28 | Baseline and day 28
  Possible scores range from 0 (Very slightly) to 6 (Very serious) 0=Very slightly 1=Slight 2=A little slightly 3=About medium 4=A bit serious 5=Severe 6=Very serious Change = (day 28 Score - Baseline Score).
Change from Baseline on the Irritable Bowel Syndrome Scale(IBS) at day 28 | Baseline and day 28
  Possible scores range from 1 (Never) to 5 (Always)
  1=Never 2=Sometimes 3=Often4=most of the time 5=Always Change = (day 28 Score - Baseline Score).

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mao R, Qiu Y, He JS, Tan JY, Li XH, Liang J, Shen J, Zhu LR, Chen Y, Iacucci M, Ng SC, Ghosh S, Chen MH. Manifestations and prognosis of gastrointestinal and liver involvement in patients with COVID-19: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2020 Jul;5(7):667-678. doi: 10.1016/S2468-1253(20)30126-6. Epub 2020 May 12. PMID 32405603
- [Result] Cheung KS, Hung IFN, Chan PPY, Lung KC, Tso E, Liu R, Ng YY, Chu MY, Chung TWH, Tam AR, Yip CCY, Leung KH, Fung AY, Zhang RR, Lin Y, Cheng HM, Zhang AJX, To KKW, Chan KH, Yuen KY, Leung WK. Gastrointestinal Manifestations of SARS-CoV-2 Infection and Virus Load in Fecal Samples From a Hong Kong Cohort: Systematic Review and Meta-analysis. Gastroenterology. 2020 Jul;159(1):81-95. doi: 10.1053/j.gastro.2020.03.065. Epub 2020 Apr 3. PMID 32251668
- [Result] Golla R, Vuyyuru SK, Kante B, Kedia S, Ahuja V. Disorders of gut-brain interaction in post-acute COVID-19 syndrome. Postgrad Med J. 2022 Jul 1:postgradmedj-2022-141749. doi: 10.1136/pmj-2022-141749. Online ahead of print. PMID 35777934
- [Result] Schmulson M, Ghoshal UC, Barbara G. Managing the Inevitable Surge of Post-COVID-19 Functional Gastrointestinal Disorders. Am J Gastroenterol. 2021 Jan 1;116(1):4-7. doi: 10.14309/ajg.0000000000001062. No abstract available. PMID 33273261
- [Result] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- [Result] Margolis KG, Cryan JF, Mayer EA. The Microbiota-Gut-Brain Axis: From Motility to Mood. Gastroenterology. 2021 Apr;160(5):1486-1501. doi: 10.1053/j.gastro.2020.10.066. Epub 2021 Jan 22. PMID 33493503
- [Result] Fan Y, Pedersen O. Gut microbiota in human metabolic health and disease. Nat Rev Microbiol. 2021 Jan;19(1):55-71. doi: 10.1038/s41579-020-0433-9. Epub 2020 Sep 4. PMID 32887946
- [Result] Zuo T, Wu X, Wen W, Lan P. Gut Microbiome Alterations in COVID-19. Genomics Proteomics Bioinformatics. 2021 Oct;19(5):679-688. doi: 10.1016/j.gpb.2021.09.004. Epub 2021 Sep 21. PMID 34560321
- [Result] Hazan S, Stollman N, Bozkurt HS, Dave S, Papoutsis AJ, Daniels J, Barrows BD, Quigley EM, Borody TJ. Lost microbes of COVID-19: Bifidobacterium, Faecalibacterium depletion and decreased microbiome diversity associated with SARS-CoV-2 infection severity. BMJ Open Gastroenterol. 2022 Apr;9(1):e000871. doi: 10.1136/bmjgast-2022-000871. PMID 35483736
- [Result] Chen Y, Gu S, Chen Y, Lu H, Shi D, Guo J, Wu WR, Yang Y, Li Y, Xu KJ, Ding C, Luo R, Huang C, Yu L, Xu M, Yi P, Liu J, Tao JJ, Zhang H, Lv L, Wang B, Sheng J, Li L. Six-month follow-up of gut microbiota richness in patients with COVID-19. Gut. 2022 Jan;71(1):222-225. doi: 10.1136/gutjnl-2021-324090. Epub 2021 Apr 8. No abstract available. PMID 33833065
- [Result] Tian Y, Sun KY, Meng TQ, Ye Z, Guo SM, Li ZM, Xiong CL, Yin Y, Li HG, Zhou LQ. Gut Microbiota May Not Be Fully Restored in Recovered COVID-19 Patients After 3-Month Recovery. Front Nutr. 2021 May 13;8:638825. doi: 10.3389/fnut.2021.638825. eCollection 2021. PMID 34055851
- [Result] Su Q, Lau RI, Liu Q, Chan FKL, Ng SC. Post-acute COVID-19 syndrome and gut dysbiosis linger beyond 1 year after SARS-CoV-2 clearance. Gut. 2023 Jun;72(6):1230-1232. doi: 10.1136/gutjnl-2022-328319. Epub 2022 Aug 8. No abstract available. PMID 35940857
- [Result] Wauters L, Ceulemans M, Schol J, Farre R, Tack J, Vanuytsel T. The Role of Leaky Gut in Functional Dyspepsia. Front Neurosci. 2022 Mar 29;16:851012. doi: 10.3389/fnins.2022.851012. eCollection 2022. PMID 35422683
- [Result] Zhou L, Zeng Y, Zhang H, Ma Y. The Role of Gastrointestinal Microbiota in Functional Dyspepsia: A Review. Front Physiol. 2022 Jun 8;13:910568. doi: 10.3389/fphys.2022.910568. eCollection 2022. PMID 35755434
- [Result] Mazzawi T. Gut Microbiota Manipulation in Irritable Bowel Syndrome. Microorganisms. 2022 Jun 30;10(7):1332. doi: 10.3390/microorganisms10071332. PMID 35889051
- [Result] Hsieh PC, Chao YC, Tsai KW, Li CH, Tzeng IS, Wu YK, Shih CY. Efficacy and Safety of Complementary Therapy With Jing Si Herbal Tea in Patients With Mild-To-Moderate COVID-19: A Prospective Cohort Study. Front Nutr. 2022 Mar 14;9:832321. doi: 10.3389/fnut.2022.832321. eCollection 2022. PMID 35369061

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT05668104/Prot_002.pdf
  • Informed Consent Form (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT05668104/ICF_003.pdf